CLINICAL TRIAL: NCT04558307
Title: Enhancing Rapid Health Response in National Crises: Feasibility of Rapid COVID-19 Testing in Disadvantaged Populations Through Community-Academic Partnerships
Brief Title: Feasibility of Rapid COVID-19 Testing in Disadvantaged Populations
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Principal Investigator, Mayo Clinic
Other Study IDs: 20-004046
Record Dates: First submitted 2020-09-18; First posted 2020-09-22 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Coronavirus Disease (COVID-19)
Keywords: COVID-19; testing; community engagement; Community-based participatory research; racial and ethnic minorities; community health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Intervention: Rapid SARS-CoV-2 testing strategy
  Interventions: Diagnostic Test: Pilot a rapid SARS-CoV-2 testing strategy
- Behavioral Intervention: Community-driven messages to promote COVID-19 testing
  Interventions: Other: Community-driven messages to promote COVID-19 testing

INTERVENTIONS:
Diagnostic Test: Pilot a rapid SARS-CoV-2 testing strategy — Rapid testing strategy at an FQHC using Mayo Clinic Laboratory (MCL) diagnostic processing with a real-time polymerase chain reaction assay for SARS-CoV-2 and a Mayo Clinic drive-through collection protocol.
  Groups: Observational Intervention
Other: Community-driven messages to promote COVID-19 testing — A one-time communication about the availability of COVID-19 testing at the FQHC to patients randomized to the intervention group using any available means of communication (text and/or mailed letter).
  Groups: Behavioral Intervention

SUMMARY:
The purpose of this study is to assess the feasibility of establishing severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) testing at a federally-qualified health center (FQHC) during a global health crisis to mitigate COVID-19 disparities in socioeconomically disadvantaged populations.

DETAILED DESCRIPTION:
Accurate and early diagnosis of COVID-19 infections are critical for rapid initiation of quarantine interventions to reduce population spread and to provide appropriate medical care to reduce related morbidity and mortality during the current pandemic. The purpose of this study is to assess the feasibility of establishing a drive-through rapid COVID-19 testing site at a federally-qualified health center (FQHC) during a global health crisis to mitigate health consequences in socioeconomically disadvantaged populations. The investigators also seek to evaluate the effectiveness of community-driven communication in increasing access to rapid testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in this population. This will inform public health decisions about improving access to testing for SARS-CoV-2 in underserved populations, particularly those receiving care in FQHCs or community health centers.

The specific aims of the study are to:

Aim 1. To determine the feasibility of a community-engaged research partnership to support rapid SARS-CoV-2 testing for symptomatic patients of all ages in the underserved population during the COVID-19 crisis. A rapid testing strategy (drive-through testing site) at a FQHC using Mayo Clinic Laboratory (MCL) diagnostic processing will be piloted.

Aim 2. To compare the effectiveness of community-driven messaging in increasing uptake of rapid SARS-CoV-2 testing compared with usual sources of health information. A simple random sample will be drawn of FQHC patients (N=1000, age 18+) with 1:1 randomization of communication about COVID-19 and availability of rapid testing from the FQHC versus usual sources (control).

ELIGIBILITY:
Inclusion Criteria:

* This study will include all patients receiving clinically indicated testing for COVID-19 at a federally qualified health center (FQHC, Open Cities Health Center, St. Paul, MN).
* There will be no formal recruitment of patients in this research.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving care at Open Cities Health Center.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility Measures - FQHC Staff | 6-months after intervention start
  FQHC staff will complete a comprehensive electronic survey adapted from the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) instrument to assess feasibility of community-engaged research partnership to support testing site (Weiner BJ, et al. Implementation Science. 2017;12(1):108.).
2. Uptake of rapid SARS-CoV-2 testing strategy at the FQHC- Effectiveness of community-driven messaging to patients | 6-months after intervention start
  Comparison of number of tests completed per group (intervention vs. control)
Uptake of rapid SARS-CoV-2 testing strategy at the FQHC | 9-months after intervention start
  Comparison of number of tests completed per group (intervention vs. control)

SECONDARY OUTCOMES:
Intervention Satisfaction Measures - Participant Satisfaction with COVID-19 testing | 6-months after intervention start
  All randomized patients will complete a comprehensive survey with questions probing satisfaction with the drive-through testing site (ease of use, process, return of results, etc.).
5. Intervention Satisfaction Measures - Participant Satisfaction with community-driven messaging | 6-months after intervention start
  Compare the satisfaction of community-driven messaging on availability of rapid SARS-CoV-2 testing at the FQHC (intervention vs. control)

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess C Brewer, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials